CLINICAL TRIAL: NCT03822975
Title: Bivalirudin With Prolonged Full Dose Infusion Versus Heparin Alone During: a Multicenter, Randomized, Open-label Trial
Brief Title: Bivalirudin With Prolonged Full Dose Infusion Versus Heparin Alone During Emergency PCI
Acronym: BRIGHT-4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shenyang Northern Hospital (Other)
Responsible Party: Principal Investigator, Han Yaling, Director, Shenyang Northern Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-031
Record Dates: First submitted 2019-01-29; First posted 2019-01-30 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: ST Elevation Myocardial Infarction
Keywords: Primary percutaneous coronary intervention; anticoagulant agents; bivalirudin; heparin
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — bivalirudin; Heparin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bivalirudin (Experimental): Bivalirudin with prolonged full dose infusion during primary PCI
  Interventions: Drug: Bivalirudin
- Heparin (Active Comparator): Heparin alone during primary PCI
  Interventions: Drug: unfractionated Heparin

INTERVENTIONS:
Drug: Bivalirudin — Bivaliruding 0.75 mg/kg intravenous bolus loading dose, and immediately followed by intravenous infusion of 1.75 mg/kg/h until 2-4 hours after PCI. It is recommended that ACT be monitored 5 minutes after the first administration, and if ACT is <225 s (Hemotec method), intravenous injection of 0.35 mg/kg of bivalirudin should be administered, and the ACT re-checked to ensure it is >225 seconds.
  Arms: Bivalirudin
Drug: unfractionated Heparin — Heparin 70 U/kg is started before coronary angiography. ACT is monitored 5 min after the first administration, and if the ACT <225 s (Hemotec method), an intravenous injection of 1000 U of heparin is administered, and the ACT re-checked to ensure it is >225 seconds.
  Arms: Heparin

SUMMARY:
This study is aimed to investigate if the bivaliruding with prolonged full dose infusion after PCI is superior to heparin alone in reducing 30-day mortality or major bleeding for patients with STEMI treated with emergency PCI. A total of 6000 STEMI patients will be enrolled and randomly assigned to receive bivalirudin or heparin during emergency PCI in a 1:1 ratio. This study will provide key evidence for peri-operative anticoagulant therapy decisions in STEMI patients.

ELIGIBILITY:
Inclusion Criteria:

* Any age;
* STEMI patients undergoing primary PCI with ST elevation≥1mm in≥2 contiguous leads or new LBBB with symptom onset 48h;
* Patients requiring staged revascularization of non-culprit vessels within 30 days may be enrolled. In such cases the same antithrombotic agents and PCI procedures must be used in the staged procedure consistent with the index procedure PCI, in particular the assigned antithrombin agent heparin vs. bivalirudin);
* Dual antiplatelet drugs must be administrated according to guidelines before PCI (loading doses and maintenance doses of aspirin and clopidogrel or ticagrelor);
* The subject or legal representative has been informed of the nature of the study, understood the provisions of the protocol, was able to ensure adherence, and signed informed consent.

Exclusion Criteria:

* Not suitable for emergency primary PCI;
* STEMI treated by thrombolysis;
* Patients received heparin, LMWH, fondaparinux, bivalirudin, or GPI within 48 hours before the index PCI;
* Mechanical complications (such as ventricular septal rupture, papillary muscle rupture with acute mitral regurgitation, etc.);
* Known allergy or contraindications to heparin, bivalirudin, aspirin, or both clopidogrel and ticagrelor
* Patients in whom the investigators consider inappropriate to participate in this study (eg, have participated in another drug/instrument study or undergoing another drug/instrument study).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6016 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2022-05-07 (Actual); Study Completion 2023-05-06 (Actual)

PRIMARY OUTCOMES:
Composite of all-cause death or BARC type 3~5 bleeding | 30 days
  BARC=Bleeding academic research consortium

SECONDARY OUTCOMES:
All cause mortality | 30 days
BARC type 3-5 bleeding | 30 days
  BARC=Bleeding academic research consortium
Major adverse cardiac and cerebral events (MACE) | 30 days
  MACE is defined as a composite of all cause death, recurrent myocardial infarction, stroke or ischemic driven target vessel revascuarlization
Net adverse clinical events (NACE) | 30 days
  NACE is defined as a composite of MACE or BARC type 3-5 bleeding
Composite of all-cause death or BARC type 2-5 bleeding | 30 days
  BARC=Bleeding academic research consortium
BARC type 2-5 bleeding | 30 days
  BARC=Bleeding academic research consortium
Stent thrombosis | 30 days
  Definite or probable stent thrombosis according to Academic Research Consortium
Thrombocytopenia | 30 days
  defined as platelet counts less than 150*10^9/L after treatment
All cause mortality | 1 years

CONTACTS AND LOCATIONS:
Overall Officials: Yaling Han, MD, Principal Investigator — The General Hospital of Northern Theater Command
Locations (85):
- China (85):
  - Bengbu Second People's Hospital, Bengbu, Anhui
  - Fu Yang People'S Hospital, Fuyang, Anhui
  - Linquan County Peoples Hospital, Fuyang, Anhui
  - NO.2 People's Hospital of Fuyang City, Fuyang, Anhui
  - Taihe County People'S Hospital, Fuyang, Anhui
  - Bozhou Peoples Hospital, Haozhou, Anhui
  - Huainan Oriental Hospital Group Affiliated Hospital of Anhui University of Science & Technology, Huainan, Anhui
  - The First Hospital of Anhui University of Science&Technology, Huainan, Anhui
  - Suzhou Municipal Hospital, Suzhou, Anhui
  - Beijing Luhe Hospital.Capital Medical University, Beijing, Beijing Municipality
  - Peking University Third Hospital Yanqing Hospital, Beijing, Beijing Municipality
  - Chongqing University Fuling Hospital, Chongqing, Chongqing Municipality
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Meizhou Peopie's Hospital, Meizhou, Guangdong
  - Yulin First People's Hospital, Yulin, Guangxi
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Affiliated Hospital Ofzunyi Medical University, Zunyi, Guizhou
  - Hengshuicardiovascularhospital, Hengshui, Hebei
  - Jiaozuo People's Hospital, Jiaozuo, Henan
  - Kaifeng Central Hospital, Kaifeng, Henan
  - Luohe Central Hospital, Luohe, Henan
  - The First People'S Hospital of Ruzhou, Ruzhou, Henan
  - Shangqiu first people's Hospital, Shangqiu, Henan
  - The Third Affiliated Hospital Of Xinxiang Medical University, Xinxiang, Henan
  - Yuzhoucitypeopleshospital, Yingchuan, Henan
  - Fuwai Central China Cardiovascular Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University Center 1, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University Center 2, Zhengzhou, Henan
  - The First People'S Hospital of Xinmi, Zhengzhou, Henan
  - Itchoshtal Tonjinee Colere Hoatono Innehatyor Seene Ano Thohholdcy, Wuhan, Hubei
  - Tongji Hospital Tongji Medical College of Hust, Wuhan, Hubei
  - Wuhanasia Heart Hospital, Wuhan, Hubei
  - Lou Di Central Hospital, Loudi, Hunan
  - Xiangtan Central Hospital, Xiangtan, Hunan
  - Yueyang Central Hospital, Yueyang, Hunan
  - Chifeng College Affiliated Hospital, Chifeng, Inner Mongolia
  - Nanjing Firsthospital, Nanjing, Jiangsu
  - Jiangsutaizhou Peoples Hospital, Taizhou, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - First Affiliated Hospital Of Gannan Medical University, Ganzhou, Jiangxi
  - Ganzhou Municipal Hospital, Ganzhou, Jiangxi
  - Nan Fang Hospital.Ganzhou, Ganzhou, Jiangxi
  - The Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - The Second Affiliated Hospital Of Nanchang University, Nanchang, Jiangxi
  - Thefirstaffiliated Hospitalofnanchang University, Nanchang, Jiangxi
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - The Second Hospital of Jilin University, Changchun, Jilin
  - Yanbian University Hospital, Yanbian, Jilin
  - General Hospital of Benxi Iron & Steel Industry Group of Liaoning Health Industry Group, Benxi, Liaoning
  - Dalian No.3 People'S Hospital, Dalian, Liaoning
  - Jiangpiqiao99@sina.com, Diaobingshancun, Liaoning
  - Fushun Central Hospital, Fushun, Liaoning
  - General Hospital of Fushun Mining Industry Group of Liaoning Health Industry Group, Fushun, Liaoning
  - General Hospital of Fuxin Mining Industry Group of Liaoning Health Industry Group, Fuxin, Liaoning
  - General Hospital of Northern Theater Command, Shenyang, Liaoning
  - The Fourth Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - The Second Hospital of Shen Yang Medical College, Shenyang, Liaoning
  - Heze Mudan People's Hospital, Heze, Shandong
  - Heze Municipal Hospital, Heze, Shandong
  - Jinan Central Hospital, Jinan, Shandong
  - Shandong Scend Provincial General Hosptial, Jinan, Shandong
  - The Fifth People's Hospital of Jinan, Jinan, Shandong
  - Qingdao Municipal Hospital, Qingdao, Shandong
  - Taian City Central Hospital, Tai’an, Shandong
  - The People's Hospital ofXin Tai City, Xintai, Shandong
  - Zao Zhuang Central Hospital Of Shandong Guoxin Healthcare Group, Zaozhuang, Shandong
  - Datong Third People'S Hospiatl, Datong, Shanxi
  - Shanxi Cardiovascular Hospital, Taiyuan, Shanxi
  - Department of Cardiology, Tangdu Hospital, Airforce Medical University, Xi’an, Shanxi
  - The Amliated HospitalofNorthwest University Xi'an No.3 Hospital, Xi’an, Shanxi
  - The Second Affiliated Hospital Of Xian Jiaotong University, Xi’an, Shanxi
  - Yan 'an university Affiliated Hospital, Yanan, Shanxi
  - The First Hospital of Liangshan, Xichang, Sichaun
  - The People's Hospital Of Pingchang, Bazhong City, Sichuan
  - "West China Hospital Sichuan University", Chengdu, Sichuan
  - Chengdu Second People'S Hospital, Chengdu, Sichuan
  - Hospital of Chengdu University of TCM, Chengdu, Sichuan
  - The Affiliated Traditional Chinese Medicine Hospital of Southwest Medical University, Luzhou, Sichuan
  - Xi Chang People'S Hospital, Xichang, Sichuan
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - The Fifth Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Yunnan St.John'S Hospital, Kunming, Yunnan
  - Zhejiang Provincial Hospital of Chinese Medicine, Hangzhou, Zhejiang
  - Taizhou Central Hospital, Taizhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li Y, Liang Z, Qin L, Wang M, Wang X, Zhang H, Liu Y, Li Y, Jia Z, Liu L, Zhang H, Luo J, Dong S, Guo J, Zhu H, Li S, Zheng H, Liu L, Wu Y, Zhong Y, Qiu M, Han Y, Stone GW. Bivalirudin plus a high-dose infusion versus heparin monotherapy in patients with ST-segment elevation myocardial infarction undergoing primary percutaneous coronary intervention: a randomised trial. Lancet. 2022 Nov 26;400(10366):1847-1857. doi: 10.1016/S0140-6736(22)01999-7. Epub 2022 Nov 6. PMID 36351459
- [Derived] Zhang D, Li Y, Qiu M, Liang Z, Xu K, Li Y, Zhang G, Xie W, Zeng H, Cheng Y, Liu J, Cheng X, Zeng Q, Zhu K, Hu J, Cheng K, Wang J, Cheng R, Zhou Y, Wang B, Cao G, Han Y, Stone GW. BMI differences on anticoagulation with bivalirudin vs. heparin during primary PCI: a BRIGHT-4 subanalysis. BMC Med. 2025 Sep 30;23(1):525. doi: 10.1186/s12916-025-04374-7. PMID 41029353
- [Derived] Su X, Qiu M, Gu C, Yang X, Liu B, Meng F, Ning B, Li W, Zhong Z, Wang Z, Shi B, Shang Z, Liang Z, Li Y, Han Y, Stone GW. Analysis of inter-hospital transfer on clinical outcomes after primary percutaneous coronary intervention for ST-segment elevation myocardial infarction: A secondary analysis of the BRIGHT-4 trial. PLoS Med. 2025 Jul 23;22(7):e1004679. doi: 10.1371/journal.pmed.1004679. eCollection 2025 Jul. PMID 40700454
- [Derived] Liao J, Qiu M, Feng X, Chen K, Zhang D, Zou Y, Zheng X, Zhao G, Tian N, Zheng Z, Peng X, Yang Q, Liang Z, Li Y, Han Y, Stone GW. Bivalirudin versus heparin in patients with or without bail-out GPI use: a pre-specified subgroup analysis from the BRIGHT-4 trial. BMC Med. 2024 Sep 27;22(1):410. doi: 10.1186/s12916-024-03579-6. PMID 39334129